CLINICAL TRIAL: NCT05110924
Title: A Large Pragmatic RCT Investigating Treatment Versus Non Treatment of Low-risk BCCs in Elderly
Brief Title: RCT Treatment Versus Non Treatment of Low-risk BCCs in Elderly
Acronym: BASINEL
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low recruitment
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: BASINEL
Record Dates: First submitted 2021-10-14; First posted 2021-11-08 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Basal Cell Carcinoma; Elderly
Keywords: Watchful waiting; Active surveillance
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: The patient will go through the stratification and randomization process and will be randomly allocated to either the treatment or the non-treatment arm of the study.
  The treatment (i.e. surgery, topical treatment or CO2-laser) will be performed by an independent dermatologist of the investigator's department who is blinded and is not aware of the patient's participation in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment arm (T-arm) (Other): Patients in the T-arm will receive diagnostic investigation(s) as in standard care. This includes clinical and dermoscopic examination and (in most cases) a biopsy to confirm the diagnosis of a BCC. Patients will be asked to fill out a questionnaire (Q) concerning their HrQoL. Important is the possible exclusion of patients (when the biopsy shows the lesion is not a BCC) in this step.
  Patients will receive treatment of their BCC in accordance with the standard treatment regimen. The treatment will be performed by an independent dermatologist of the investigator's department who is blinded and not aware of the patient's participation in this study. After the treatment, a new Q will be sent out to capture the HrQoL and possible patient-reported side effects. Afterwards, the patients will be followed every 6 to 12 months for 36 months with a clinical evaluation of the previously treated skin site, evaluation of possible complications and the HrQoL and complications Qs.
  Interventions: Other: Standard of care
- non-Treatment arm (n-T-arm) (Other): Patients allocated to the n-T-arm will receive diagnostic investigations by non-invasive imaging techniques to confirm the diagnosis of a BCC. Patients will be asked to fill out a Q concerning their HrQoL. Important to point out is the possible exclusion of certain patients (when the imaging shows the lesion is not a BCC) in this step.
  The patients in this arm will be followed every 6 to 12 months for 36 months. Every study visit there will be a clinical evaluation of the tumor. At the follow-up visits of 6, 12, 24 and 36 months a new documentation of the tumor will take place with in vivo imaging. At these time-points, patients will also be asked to fill out the HrQoL Q and complications Q.
  Because of ethical reasons, a maximum tolerable diameter of the tumor has been defined in advance: BCCs in the non-treatment arm that reach a diameter of 4cm will be excluded and will receive treatment.
  Interventions: Other: Monitoring

INTERVENTIONS:
Other: Standard of care — Patients in the treatment arm will receive standard care.
  Arms: Treatment arm (T-arm)
Other: Monitoring — Patients in the non-treatment arm will be closely monitored: the tumor will be evaluated using non-invasive imaging devices based on multispectral dermoscopy, reflectance confocal microscopy to determine the exact histology and high definition optical coherence tomography for imaging and volume calculation of the BCC.
  Arms: non-Treatment arm (n-T-arm)

SUMMARY:
This study will be a randomized controlled trial (RCT). Patients with a minimum age of 75 years who consult at the dermatology department of the Ghent University Hospital and who are diagnosed with minimum one lesion suspicious for a low-risk basal cell carcinoma will be asked to participate in this study.

Rationale: Basal cell carcinomas (BCCs) represent 70% of all skin cancers. These tumors do not metastasize but are locally invasive if left untreated. There is a high incidence of BCC in elderly and clinicians frequently face important treatment dilemmas. The approach to BCC in elderly should be investigated thoroughly, since current data on health-related quality of life, complication risks and biological behavior of these tumors is absent, and most guidelines are based on studies in young patients.

Objective: The investigators will examine the possibility of not treating all BCCs by collecting data on the in vivo biological behavior of low-risk basal cell carcinomas in elderly patients with state-of-the-art imaging techniques. The investigators want to combine tumor characteristics with patient profiles, in order to estimate whether a chosen treatment will positively affect the patients' quality of life within a predetermined timeframe.

Study design: Randomized controlled trial (RCT) with study visits every 6 to 12 months for a total follow-up period of 36 months.

Study population: Patients consulting at the Department of Dermatology of the Ghent University Hospital with the minimum age of 75 years and a new diagnosis of (a) low-risk basal cell carcinoma(s).

Intervention: Evaluation of the impact on the quality of life and the complication risks in both study arms. In addition, survival data will be gathered in both study arms. In the non-treatment arm, there will be an evaluation of the biological behavior of these low-risk basal cell carcinomas using in vivo imaging devices.

Patients in the treatment arm will receive standard care. Patients in the non-treatment arm will be closely monitored: the tumor will be evaluated using non-invasive imaging devices. Patients will be asked to fill in a questionnaire concerning their HrQoL at consecutive time points. Also patient-reported side effects will be evaluated via a questionnaire. The investigators will compare standard treatment versus non-treatment (1:1 allocation) in a randomized controlled trial.

Subjects can withdraw from participating in this study at any time for any reason without any consequences.

DETAILED DESCRIPTION:
See protocol

ELIGIBILITY:
Inclusion Criteria:

- Patients with the age of 75 years or older with a new diagnosis of at least one basal cell carcinoma localized on the trunk or on the limbs (with the exception of BCCs on the hands and/or the feet).

Exclusion Criteria:

* Patient is unable to provide consent.
* Patient is unable to understand the task and questionnaires.
* Patient is immunocompromised.
* Patient has a genetic skin cancer syndrome.
* The BCC has a diameter of more than 3 cm.
* The BCC occurs in a skin site that underwent radiotherapy in the past.
* Patient is being treated with chemoprevention for KC or underwent a recent field treatment for KC in the region of the low-risk BCC.
* Patient has a history of malignant melanoma or other types of NMSC (with the exception of KC).
* Patient has had a high-risk SCC during the last 2 years or a SCC in the head and neck region during the last 2 years.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Health-related Quality of Life | Day 0
  To determine the impact on the health-related quality of life in elderly patients with low-risk basal cell carcinomas in the treatment versus the non-treatment arm.
Health-related Quality of Life | Day of Treatment
  To determine the impact on the health-related quality of life in elderly patients with low-risk basal cell carcinomas in the treatment versus the non-treatment arm.
Health-related Quality of Life | Month 6
  To determine the impact on the health-related quality of life in elderly patients with low-risk basal cell carcinomas in the treatment versus the non-treatment arm.
Health-related Quality of Life | Month 12
  To determine the impact on the health-related quality of life in elderly patients with low-risk basal cell carcinomas in the treatment versus the non-treatment arm.
Health-related Quality of Life | Month 24
  To determine the impact on the health-related quality of life in elderly patients with low-risk basal cell carcinomas in the treatment versus the non-treatment arm.
Health-related Quality of Life | Month 36
  To determine the impact on the health-related quality of life in elderly patients with low-risk basal cell carcinomas in the treatment versus the non-treatment arm.
Complication risks | Day of Treatment
  To determine the complication risk in elderly patients with low-risk basal cell carcinomas in the treatment versus the non-treatment arm.
Complication risks | Month 6
  To determine the complication risk in elderly patients with low-risk basal cell carcinomas in the treatment versus the non-treatment arm.
Complication risks | Month 12
  To determine the complication risk in elderly patients with low-risk basal cell carcinomas in the treatment versus the non-treatment arm.
Complication risks | Month 24
  To determine the complication risk in elderly patients with low-risk basal cell carcinomas in the treatment versus the non-treatment arm.
Complication risks | Month 36
  To determine the complication risk in elderly patients with low-risk basal cell carcinomas in the treatment versus the non-treatment arm.

SECONDARY OUTCOMES:
Survival | Month 36 + 10 years
  To determine the survival of elderly patients with low-risk basal cell carcinoma in the treatment versus the non-treatment arm.
Natural behavior | Day 0
  To evaluate the in vivo natural behavior and growth of the basal cell carcinomas in the non-treatment arm.
Natural behavior | Month 6
  To evaluate the in vivo natural behavior and growth of the basal cell carcinomas in the non-treatment arm.
Natural behavior | Month 12
  To evaluate the in vivo natural behavior and growth of the basal cell carcinomas in the non-treatment arm.
Natural behavior | Month 24
  To evaluate the in vivo natural behavior and growth of the basal cell carcinomas in the non-treatment arm.
Natural behavior | Month 36
  To evaluate the in vivo natural behavior and growth of the basal cell carcinomas in the non-treatment arm.

OTHER OUTCOMES:
Treatment effectiveness | Month 36
  To determine treatment effectiveness (recurrence rates of the BCCs after 36 months) of the different (standard of care) therapies administered in the treatment arm.

CONTACTS AND LOCATIONS:
Overall Officials: Lieve Brochez, MD, PhD, Principal Investigator — Ghent University Hospital, Department of Dermatology
Locations (1):
- Department of Dermatology, Ghent University Hospital, Ghent, East Flanders, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Van Coile L, Verhaeghe E, Ongenae K, Brochez L, Hoorens I. Study protocol of the BASINEL Study: a pragmatic randomised controlled trial investigating treatment versus no treatment of low-risk basal cell carcinomas in older persons. BMJ Open. 2022 Nov 10;12(11):e063526. doi: 10.1136/bmjopen-2022-063526. PMID 36356999